CLINICAL TRIAL: NCT05474092
Title: Evaluation of the Aeson® Total Artificial Heart (TAH) System in a Post-Market Approval Setting
Brief Title: Aeson TAH System - Post-Market Clinical Follow-up Study
Status: Recruiting | Type: Observational
Sponsor: Carmat SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: CAR2021-PM
Record Dates: First submitted 2021-06-29; First posted 2022-07-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: Advanced Heart Failure; Total Artificial Heart; Bridge to Transplant
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Aeson Total Artificial Heart — Heart Replacement Therapy

SUMMARY:
The safety and performance of the Aeson TAH system have been demonstrated for the CE mark approval in December 2020. The purpose of this post-market clinical investigation is to confirm the safety, performance and effectiveness of the Aeson TAH system when used in routine care by surgeons.

DETAILED DESCRIPTION:
The Primary objective/endpoint is survival rate on the originally implanted Aeson device at 90 days post-implant (H1 > 64%).

The second objectives/endpoints are:

1. Confirm the performance and safety profile of the device for patients implanted with the Aeson TAH system until being transplanted:

   * Survival at 6, 12, 18, and 24-months post-implant, and total support duration before transplantation;
   * Health status change as measured by NYHA classification, 6MWT and Quality of Life Questionnaire (EQ-5D-5L);
   * Renal and hepatic function as measured by biological parameters;
   * Hemocompatibility profile measured by biological parameters and incidence of hemocompatible-related adverse events;
   * Frequency and Incidence of Serious Adverse events.
2. Assess the effectiveness of device upgrades
3. Confirm the safety profile of the device for patients after being transplanted.

   * Survival at 30 days, 6 months, and 12 months post-transplant
   * Frequency and Incidence of Serious Adverse Event of special interest as graft reject, neurological events, major bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patient is intended to receive an Aeson TAH system according to the IFU indications within standard medical practice
* Patient has provided written informed consent using the Ethics Committee approved consent form

Non-inclusion Criteria:

* Vulnerable populations who could not voluntarily consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients intended to receive Aeson TAH system as per commercial use
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 90 days post-implant
  Proportion of patients surviving on the originally implanted Aeson device (superiority test > 64%)

SECONDARY OUTCOMES:
Survival and total support duration before transplantation | 6, 12, 18 and 24-months post-implant
  Survival post-implant
Health status change before transplantation | 3, 6, 9, 12, 18 and 24-months post-implant
  Measured by EuroQol EQ-5D-5L questionnaire, health-related quality of life consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses (EQ-5D-5L). The responses record five levels of severity (1:no problems; 2:slight problems; 3:moderate problems 4:severe problems; 5:extreme problems) within a particular EQ-5D dimension
Functional status change before transplantation | 3, 6, 9, 12, 18 and 24-months post-implant
  Measured by 6 minutes walking distance in meters
Length of hospital stay and time at home before transplantation | 3, 6, 9, 12, 18 and 24-months post-implant
  Measured with discharge timing, frequency and duration of rehospitalizations; time at home or rehabilitation site
Frequency and Incidence of Serious Adverse events before transplantation | 3, 6, 9, 12, 18 and 24-months post-implant
  As defined by INTERMACS
Assess the effectiveness of device upgrades | Between 3 and 24 months post-implantation, when heart transplant occurred
  Standard expertise of explanted device
Confirm the safety profile of the device after transplantation | 30 days, 3 months, 6 months, 12 months post-transplantation
  Survival after transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- HZ Dresden, Dresden, Germany